CLINICAL TRIAL: NCT01877005
Title: A Phase II Study of Oral JAK1/JAK2 Inhibitor INC424 in Adult Patients With Relapsed/Refractory Classical Hodgkin's Lymphoma
Acronym: HIJAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIJAK
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Hodgkin's Lymphoma
Keywords: Multicenter, single arm and opened label phase II study
MeSH Terms: conditions — Hodgkin Disease | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolitinib (Experimental): Induction period: Ruxolitinib will be given twice daily during 6 cycles of 28 days.
  Maintenance period: patients who achieve at least a stable disease (according Cheson 2007) at the end of cycle 6 and for whose a clinical benefit is observed according to the Investigator's opinion will be eligible for maintenance treatment by ruxolitinib twice daily every day of 28-day cycles.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib
  Other Names: JAKAVI

SUMMARY:
Phase II study to assess the efficacy of 6 cycles of oral JAK1/2 inhibitor ruxolitinib in patients with advanced Hodgkin's lymphoma for whom no curative option is available.

ELIGIBILITY:
Inclusion critera:

* Patients ≥ 18 years with classical HL relapsing or refractory after at least 1 prior systemic therapy. Patients must have relapsed after high-dose therapy with ASCT, or have been deemed ineligible for high-dose therapy with ASCT
* ECOG performance status ≤ 3
* Measurable nodal disease: 1 cm in the longest transverse diameter and clearly measurable in at least two perpendicular dimensions, as determined by CT scan (MRI is allowed only if CT scan cannot be performed).
* Patient has the following laboratory values:

  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L [SI units 1.0 x 10^9/L]
  * Platelet count ≥ 75 x 10^9/L]
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Serum bilirubin ≤ 1.5 x ULN (or ≤ 3.0 x ULN, if patient has Gilbert syndrome)
  * AST/SGOT and/or ALT/SGPT ≤ 2.5 x ULN or ≤ 5.0 x ULN if the transaminase elevation is due to liver disease involvement
* Signed written informed consent
* Life expectancy ≥ 3 months
* Corrected QT interval ≤ 450 mSec
* Men and women of childbearing potential must agree to use an adequate method of contraception during the study treatment and for at least 1 week after the last study drug administration
* The patient must be covered by a social security system (for inclusions in France)

Exclusion criteria:

* Previous treatment with ruxolitinib or another JAK inhibitor
* Contraindication to ruxolitinib
* Patient received chemotherapy or radiotherapy or any investigational drug within 14 days prior to starting study drug or whose side effects of such therapy have not resolved to ≤ grade 1
* Patient treated with allogeneic hematopoietic stem cell transplant who is currently on, or has received immunosuppressive therapy within 90 days prior to start of screening and/or have ≥ Grade 2 graft versus host disease (GvHD).
* Patient with prior history of another active primary malignancy ≤ 2 years before study entry, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix
* Any serious active disease or co-morbid medical condition that, according to the investigator's decision, will substantially increase the risk associated with the subject's participation in the study.
* Uncontrolled infectious disease, including active HBV infection defined by either detection of HBs Antigen or presence of anti HBc antibody without detectable anti HBs antibody.
* HIV, HCV or HTLV serology positivity and/or documented infection with active hepatitis B
* Prior history of CNS involvement with lymphoma
* Pregnant or lactating woman
* Adult patient unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-07-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Overall response Rate (ORR) according to Cheson 2007 | 6 months
  Overall Response Rate according to the International Working Group criteria (Cheson 2007) is defined as patient with Complete response or Partial response.
  Patient without response assessment (due to whatever reason) will be considered as non responder.

SECONDARY OUTCOMES:
Overall response rate (ORR) according to Cheson 1999 | 6 months
  Overall Response Rate according to the International Working Group criteria (Cheson 1999) is defined as patient with Complete response, unconfirmed Complete response or Partial response.
  Patient without response assessment (due to whatever reason) will be considered as non responder.
Complete response rates (CR) according to Cheson 2007 and 1999 | 2 months, 4 months and 6 months
  Assessment of response will be based on the International Workshop to Standardize Response criteria for lymphoma: Cheson, 1999 and 2007.
  Patient without response assessment (due to whatever reason) will be considered as nonresponder.
Best Response Rate (BRR) according to Cheson 1999 and 2007 | 6 months
  Disease response evaluation at 2; 4 and 6 months will be used to determine the Best Response Rate, according to Cheson 1999 and 2007.
  The Best Complete Response and Best Overall Response will be presented. Patient without response assessment (due to whatever reason) will be considered as nonresponder.
Safety endpoints | 30 months
  Description of all adverse events, vital signs measurements, clinical laboratory measurements and concomitant medications.
Time to response | Up to 30 months
  Time to response will be defined as the time from inclusion into the study to the time of attainment of PR or CR according to Cheson 2007 criteria.
Duration of response | Up to 4.5 years
  Duration of response will be measured from the time of attainment of CR or PR according to Cheson 2007 cirteria to the date of first documented disease progression, relapse or death from any cause.
  Patients alive and free of progression will be censored at their last follow-up date.
Progression Free Survival (PFS) | Up to 4.5 years
  PFS is defined at the time from inclusion into the study to the first observation of documented disease progression/relapse according to Cheson 2007 criteria or death due to any cause.
  If a subject has not progressed or died, PFS will be censored at the time of last visit.
Overall Survival (OS) | Up to 4.5 years
  OS will be measured from the date of inclusion to the date of death from any cause.
  Patients who did not died will be censored at the time of last visit.
Evaluation of systemic symptoms | Up to 30 months
  Evaluation of efficacy of ruxolitinib on systemic symptoms such as fever, sweating, fatigue and itching will be done via systemic symptoms Questionnaire designed for this purpose and completed at Baseline and then at Day1 of each visit during Induction and Maintenance period of the study

OTHER OUTCOMES:
Anatomopahtological study | baseline
  * FISH: JAK2 copies and rearrangements
  * Immunohistochemistry: JAK2 overexpression

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Den Neste, MD, Principal Investigator — Lymphoma Study Association; Franck Morschhauser, MD, Principal Investigator — Lymphoma Study Association
Locations (10):
- Belgium (2):
  - UCL Louvain St Luc, Brussels
  - Université Catholique de Louvain Mont Godinne, Yvoir
- France (8):
  - Chu Cote de Nacre, Caen
  - Hopital Henri Mondor, Créteil
  - Chu Dijon, Dijon
  - Chru de Lille, Lille
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Lyon Sud, Lyon
  - CHU de Nantes, Hotel Dieu, Nantes
  - Centre Henri Becquerel, Rouen

REFERENCES:
- [Derived] Van Den Neste E, Andre M, Gastinne T, Stamatoullas A, Haioun C, Belhabri A, Reman O, Casasnovas O, Ghesquieres H, Verhoef G, Claessen MJ, Poirel HA, Copin MC, Dubois R, Vandenberghe P, Stoian IA, Cottereau AS, Bailly S, Knoops L, Morschhauser F. A phase II study of the oral JAK1/JAK2 inhibitor ruxolitinib in advanced relapsed/refractory Hodgkin lymphoma. Haematologica. 2018 May;103(5):840-848. doi: 10.3324/haematol.2017.180554. Epub 2018 Jan 19. PMID 29351986
- See also: LYSA (the Lymphoma Study Association) — http://lysa-lymphoma.org